CLINICAL TRIAL: NCT02059408
Title: Can a Targeted Screen-and-treat Program for Chronic Kidney Disease Improve Blood Pressure (BP) Management Among Persons at High Risk for Complications ?
Brief Title: Screen-and-treat Program for Chronic Kidney Disease- High Risk Persons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP2014R34
Record Dates: First submitted 2014-01-17; First posted 2014-02-11 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care (No Intervention): The patients in this arm will receive normal primary care.
- Screen-Educate (Active Comparator): Education program to improve blood pressure control among hypertensive non-diabetic persons. The Screen and Educate arm recommends using creatinine, cystatin C and albuminuria for detection and risk stratification, followed by guideline-concordant CKD management appropriate for CKD stage.
  Interventions: Other: Screen-Educate
- Screen-Educate and Intensify Treatment (Active Comparator): Education and treatment program to improve blood pressure control among hypertensive non-diabetic persons. The Screen-Educate and Intensify Treatment adds a pharmacist-led CKD management program and attempts to improve BP management and patient-centered outcomes among persons with newly stratified higher risk CKD based on creatinine, cystatin c and albuminuria.
  Interventions: Other: Screen-Educate; Other: Screen-Educate and Intensify Treatment

INTERVENTIONS:
Other: Screen-Educate — Education program to improve blood pressure control among hypertensive non-diabetic persons. The Screen and Educate arm will recommend using creatinine, cystatin C and albuminuria for screening and risk stratification, followed by guideline-concordant CKD management appropriate for CKD stage. Recommendations are sent to the primary care provider via an electronic note.
  Arms: Screen-Educate; Screen-Educate and Intensify Treatment
Other: Screen-Educate and Intensify Treatment — This arm adds option of a pharmacist. PCPs randomized to this arm will have the additional option to refer their higher-risk patients to a clinical pharmacist-led CKD management program with education. A primary care clinical pharmacist will schedule a series of appointments with patients found to have confirmed higher-risk CKD (defined as eGFRcreat-cys <45, or eGFR 45-59 and ACR ≥ 30 mg/g). The pharmacist will follow treatment algorithms recommended by the 2012 KDIGO international CKD guidelines, and designed by a team of internists and nephrologists.
  Arms: Screen-Educate and Intensify Treatment

SUMMARY:
The overall hypothesis of this trial is that screening for chronic kidney disease, followed by education or treatment program will improve blood pressure control among hypertensive non-diabetic persons.

DETAILED DESCRIPTION:
To evaluate a CKD screen-and-educate program in primary care for improving blood pressure management compared with usual care, among non-diabetic adults with hypertension.

ELIGIBILITY:
Inclusion Criteria:

The entire primary care medical practice at SFVAMC will be considered. Randomization will occur at the team (nurse) level. Within each team, individual patients will be considered eligible for chronic kidney disease screening by this protocol and inclusion in our trial if they have hypertension without concomitant diabetes, and no prior recorded diagnosis of chronic kidney disease. Hypertension will be defined as systolic blood pressure >140 or diastolic blood pressure >90 mmHg at more than two encounters (any encounter) within the previous 3 years or a documented diagnosis of hypertension (listed in problem list or ICD-9 code). Diagnosed chronic kidney disease will be defined as a documentation of chronic kidney disease in the problem list or ICD-9 code or on-going nephrology follow up. We define diagnosed chronic kidney disease without consideration of estimated glomerular filtration rate by creatinine or albumin-creatinine-ratio in the laboratory section of the medical record, since work from our group and others has shown that awareness and recognition of chronic kidney disease is extremely low, even among persons with documented reduced estimated glomerular filtration rate or albuminuria. Persons will be required to have seen their physician at least one time within the past 18 months.

Exclusion Criteria:

Kidney transplant recipients, pregnant women, and individuals with an estimated glomerular filtration rate <15 ml/min/1.73 m2 will be excluded from this study as they likely need specialty care for uncontrolled hypertension. Persons aged >80 will be excluded because data on aggressive blood pressure lowering in this population are less clear and adverse effects associated with aggressive blood pressure control have been well documented. We will exclude persons with New York Heart Association class III or IV heart failure, known ejection fraction <25%, or documented allergy to Angiotensin-Converting Enzyme/Angiotensin II Receptor Blockers. Other exclusion criteria relate to the required ability to communicate with providers and provide informed consent: prevalent dementia, impaired cognition or severe mental illness; expected life expectancy <6 months; severe visual impairment in the absence of an available caretaker who can read.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1819 (Actual)
Dates: Start 2015-09; Primary Completion 2017-01 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen A Peralta, MD, MAS, Principal Investigator — San Francisco Veterans Affairs Medical Center; Erica Day, MPH, Study Director — San Francisco Veterans Affairs Medical Center
Locations (1):
- San Francisco Veteran Affairs Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
There is not currently a plan to make the IDP data available.

REFERENCES:
- [Background] Coresh J, Byrd-Holt D, Astor BC, Briggs JP, Eggers PW, Lacher DA, Hostetter TH. Chronic kidney disease awareness, prevalence, and trends among U.S. adults, 1999 to 2000. J Am Soc Nephrol. 2005 Jan;16(1):180-8. doi: 10.1681/ASN.2004070539. Epub 2004 Nov 24. PMID 15563563
- [Background] Peralta CA, Shlipak MG, Judd S, Cushman M, McClellan W, Zakai NA, Safford MM, Zhang X, Muntner P, Warnock D. Detection of chronic kidney disease with creatinine, cystatin C, and urine albumin-to-creatinine ratio and association with progression to end-stage renal disease and mortality. JAMA. 2011 Apr 20;305(15):1545-52. doi: 10.1001/jama.2011.468. Epub 2011 Apr 11. PMID 21482744
- [Background] Shlipak MG, Coresh J, Gansevoort RT. Cystatin C versus creatinine for kidney function-based risk. N Engl J Med. 2013 Dec 19;369(25):2459. doi: 10.1056/NEJMc1312801. No abstract available. PMID 24350959
- [Background] Stevens PE, Levin A; Kidney Disease: Improving Global Outcomes Chronic Kidney Disease Guideline Development Work Group Members. Evaluation and management of chronic kidney disease: synopsis of the kidney disease: improving global outcomes 2012 clinical practice guideline. Ann Intern Med. 2013 Jun 4;158(11):825-30. doi: 10.7326/0003-4819-158-11-201306040-00007. PMID 23732715
- [Derived] Peralta CA, Frigaard M, Rubinsky AD, Rolon L, Lo L, Voora S, Seal K, Tuot D, Chao S, Lui K, Chiao P, Powe N, Shlipak M. Implementation of a pragmatic randomized trial of screening for chronic kidney disease to improve care among non-diabetic hypertensive veterans. BMC Nephrol. 2017 Apr 12;18(1):132. doi: 10.1186/s12882-017-0541-6. PMID 28399844

RESULTS

PARTICIPANT FLOW:
Groups:
- Screen-Educate and Intensify Treatment: The Screen-Educate and Intensify Treatment adds a pharmacist-led CKD management program and attempts to improve BP management and patient-centered outcomes among persons with newly stratified higher risk CKD based on creatinine, cystatin c and albuminuria.
Period: Overall Study
Arm/Group | Usual Care | Screen-Educate | Screen-Educate and Intensify Treatment
Started | 604 | 599 | 616
Completed | 604 | 269 | 258
Not Completed | 0 | 330 | 358
Not completed — Did not get tested | 0 | 330 | 358

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Screen-Educate | Screen-Educate and Intensify Treatment | Total
Number analyzed (Participants) | 604 | 599 | 616 | 1819
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [61 to 72] | 68 [62 to 72] | 68 [61 to 72] | 68 [61 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 6 | 8
  Male | 603 | 598 | 610 | 1811
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 5 | 4 | 11
  Asian | 52 | 48 | 50 | 150
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 87 | 107 | 104 | 298
  White | 344 | 329 | 336 | 1009
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 119 | 110 | 122 | 351
Region of Enrollment [Number; unit: participants]
  United States | 604 | 599 | 616 | 1819

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Pressure
Description: Change in blood pressure from enrollment to the end of the 12-month follow up period as a continuous outcome,
Time Frame: baseline, 12 months
Measure: Median (Inter-Quartile Range); unit: mmHg
Groups:
- Screen-Educate: Education program to improve blood pressure control among hypertensive non-diabetic persons. The Screen and Educate arm recommends using creatinine, cystatin C and albuminuria for detection and risk stratification, followed by guideline-concordant chronic kidney disease (CKD) management appropriate for CKD stage.
  Screen-Educate: Education program to improve blood pressure control among hypertensive non-diabetic persons. The Screen and Educate arm will recommend using creatinine, cystatin C and albuminuria for screening and risk stratification, followed by guideline-concordant CKD management appropriate for CKD stage. Recommendations are sent to the primary care provider via an electronic note.
- Screen-Educate and Intensify Treatment: Screen-Educate and Intensify Treatment: Adds option of a pharmacist to what is described in the Screen-Educate arm. primary care physician (PCPs) randomized to this arm will have the additional option to refer their higher-risk patients to a clinical pharmacist-led CKD management program with education.
Arm/Group | Usual Care | Screen-Educate | Screen-Educate and Intensify Treatment
Number analyzed (Participants) | 604 | 599 | 616
mmHg
  Change in SBP | -1 [-11 to 11] | -2 [-11 to 11] | -2 [-13 to 10]
  Change in DBP | -2 [-7 to 4] | -2 [-7 to 4] | -1 [-7 to 5]

2. Secondary Outcome: ACE/ARB Prescription by a Clinician
Description: New use by end of the study
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Screen-Educate and Intensify Treatment: Screen-Educate and Intensify Treatment: Adds option of a pharmacist to what is described in the Screen-Educate arm. PCPs randomized to this arm will have the additional option to refer their higher-risk patients to a clinical pharmacist-led CKD management program with education.
Arm/Group | Usual Care | Screen-Educate | Screen-Educate and Intensify Treatment
Number analyzed (Participants) | 604 | 599 | 616
Participants | 26 | 38 | 39

3. Other Pre Specified Outcome: Testing Time
Description: Time in minutes to order and interpret tests. Reported by Primary Care Providers and pharmacists.
Time Frame: 24 months
Population: Data were not collected for this outcome. It was not feasible.
Arm/Group | Usual Care | Screen-Educate | Screen-Educate and Intensify Treatment
Number analyzed (Participants) | 0 | 0 | 0

4. Other Pre Specified Outcome: Testing Cost
Description: Reported by Primary Care Providers and pharmacists. Cost in dollars of testing and pharmacist time.
Time Frame: 24 months
Population: Not feasible to collect data for this outcome.
Groups:
- Screen-Educate and Intensify Treatment: Screen-Educate and Intensify Treatment: Adds option of a pharmacist to what is described in the Screen-Educate arm. Primary care physicians (PCPs) randomized to this arm will have the additional option to refer their higher-risk patients to a clinical pharmacist-led CKD management program with education.
Arm/Group | Usual Care | Screen-Educate | Screen-Educate and Intensify Treatment
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Screen-Educate and Intensify Treatment: Education and treatment program to improve blood pressure control among hypertensive non-diabetic persons. The Screen-Educate and Intensify Treatment adds a pharmacist-led CKD management program and attempts to improve BP management and patient-centered outcomes among persons with newly stratified higher risk CKD based on creatinine, cystatin c and albuminuria.
  Screen-Educate: Education program to improve blood pressure control among hypertensive non-diabetic persons. The Screen and Educate arm will recommend using creatinine, cystatin C and albuminuria for screening and risk stratification, followed by guideline-concordant CKD management appropriate for CKD stage. Recommendations are sent to the primary care provider via an electronic note.
  Screen-Educate and Intensify Treatment: Adds option of a pharmacist. PCPs randomized to this arm will have the additional option to refer their higher-risk patients to a clinical pharmacist-led CKD management program with education.
Arm/Group | Usual Care | Screen-Educate | Screen-Educate and Intensify Treatment
All-Cause Mortality (participants affected / at risk) | 0/604 | 0/599 | 0/616
Serious Adverse Events (participants affected / at risk) | 0/604 | 0/599 | 0/616
Other Adverse Events (participants affected / at risk) | 0/604 | 0/599 | 0/616

LIMITATIONS AND CAVEATS:
A limitation in this study was that over 50% of eligible patients were not tested.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT02059408/Prot_SAP_000.pdf